CLINICAL TRIAL: NCT06780930
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo- Controlled Study of Vorasidenib (S095032/AG-881) in Asian Participants With Residual or Recurrent Grade 2 Glioma With an IDH1 or IDH2 Mutation
Brief Title: Phase 3 Study of Vorasidenib (S095032/AG-881) in Asian Participants With Residual or Recurrent Grade 2 Glioma With an IDH1 orIDH2 Mutation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL3-95032-016
Record Dates: First submitted 2024-12-24; First posted 2025-01-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Residual or Recurrent Grade 2 IDH Mutant Glioma
MeSH Terms: interventions — vorasidenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized Double-Blind Phase: Vorasidenib (Experimental)
  Interventions: Drug: Vorasidenib
- Randomized Double-Blind Phase: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vorasidenib — For oral administration once daily
  Arms: Randomized Double-Blind Phase: Vorasidenib
Drug: Placebo — For oral administration once daily
  Arms: Randomized Double-Blind Phase: Placebo

SUMMARY:
The objective of this study is to determine the efficacy, safety, and pharmacokinetics of vorasidenib in Asian participants with residual or recurrent Grade 2 glioma with an IDH1 or IDH2 mutation. The study will begin with a safety lead-in (SLI) phase and then will transition to a randomized double-blind placebo-controlled phase. During the study participants will have study visits on day 1 and 15 of the first two cycles, and then only on day 1 of treatment cycles in the frequency included in the study schedule of assessments. All participants will have an end of treatment visit within 7 days after their last dose of study treatment. Approximately 28 (+5) days after treatment has ended, a safety follow-up visit will occur. Study visits may include questionnaires, blood tests, ECG, vital signs, and a physical examination. Beginning at the end of treatment visit participants will be contacted by phone every 6 months for overall survival up to 5 years after the last participant is randomized or until death, withdrawal of consent from overall study participation, lost to follow-up, or sponsor ending the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 12 years of age (for Randomized Double-Blind phase) and weigh at least 40 kg.
* Have a Karnofsky Performance Scale (KPS) score (for participants ≥16 years of age) or Lansky Play Performance Scale (LPPS) score (for participants <16 years of age) of ≥80%.
* Have Grade 2 oligodendroglioma or astrocytoma per WHO 2016 criteria.
* Have had at least 1 prior surgery for glioma with the most recent one having occurred at least 1 year (-1 month) and not more than 5 years (+3 months) before randomization, and no other prior anticancer therapy, including radiotherapy and not be in need of immediate chemotherapy or radiotherapy.
* Have confirmed IDH1 (IDH1 R132H/C/G/S/L mutation variants tested) or IDH2 (IDH2 R172K/M/W/S/G mutation variants tested) gene mutation status disease
* Have MRI-evaluable, measurable, non-enhancing disease, as confirmed by the BIRC for double blind part.

Exclusion Criteria:

* Have had any prior anticancer therapy other than surgery (biopsy, sub-total resection, gross-total resection) for treatment of glioma including systemic chemotherapy, radiotherapy, vaccines, small-molecules, IDH inhibitors, investigational agents, laser ablation, etc.
* Concurrent active malignancy except for a) curatively resected nonmelanoma skin cancer or b) curatively treated carcinoma in situ. Participants with previously treated malignancies are eligible provided they have been disease-free for 3 years at Screening.
* Have any other acute or chronic medical or psychiatric condition that may increase the risk associated with the study participation or investigational product administration or may interfere with the interpretation of study results.
* Have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, known positive human immunodeficiency virus antibody results, or AIDS-related illness. Participants with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Participants with chronic HBV that is adequately suppressed by institutional practice will be permitted.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Approximately 1.5 years
  The time from date of randomization to date of first documented radiographic progressive disease (PD), as assessed by the Blinded Independent Review Committee (BIRC), or date of death due to any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Dose limiting toxicities (DLTs) (for open-label Safety Lead In (SLI) phase) | Through Cycle 1 (28 days)
Number of adverse events (AEs), serious adverse events (SAEs), and AEs leading to discontinuation or death | Through the safety follow up visit, 28 days after the last dose (approximately 6.5 years)
Severity of AEs | Through the safety follow up visit, 28 days after the last dose (approximately 6.5 years)
Time-To-Next-Intervention (TTNI) | Through the PFS Follow-up (approximately 6.5 years)
  The time from randomization to the initiation of the first subsequent anticancer therapy (including vorasidenib, for participants randomized to placebo who subsequently cross over) or death due to any cause.
Tumor Growth Rate (TGR) as assessed by volume | Through the PFS Follow-up (approximately 6.5 years)
  Defined as the percentage change in tumor volume every 6 months
Objective response | Through the PFS Follow-up (approximately 6.5 years)
  Best overall response of Complete Response (CR), Partial Response (PR), or Minor Response (MR)
Time to response | Through the PFS Follow-up (approximately 6.5 years)
  The time from the date of randomization to the date of first documented CR, PR, or MR for responders as assessed by the Investigator and by the BIRC
Duration of response | Through the PFS Follow-up (approximately 6.5 years)
  The time from the date of first documented CR, PR, or MR to the earlier of the date of death due to any cause or first documented radiographic PD as assessed by the Investigator and by the BIRC
Overall survival | Through the Overall Survival Follow-up (approximately 6.5 years)
  The time from the date of randomization to the date of death due to any cause
Plasma concentrations of vorasidenib | Through the end of treatment visit, within 7 days after the last dose (approximately 6.5 years)
Number of seizures by month | Through the end of treatment visit, within 7 days after the last dose (approximately 6.5 years)

CONTACTS AND LOCATIONS:
Locations (8):
- China (6):
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tiantan Hospital, Beijing
  - Sanbo Brain Hospital, Capital Medical University, Beijing
  - Huashan Hospital Fudan University, Shanghai
  - The Second Affiliated Hospital of Air Force Military Medical University, Xi'an
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital,, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/